CLINICAL TRIAL: NCT05351723
Title: Effectiveness of Non-pharmacological Interventions for Dementia Among Elderly in Hai Duong Province, Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: National Geriatric Hospital (Other Government)
Responsible Party: Principal Investigator, Vu Thu Huong, MD, Principal Investigator, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #HMUIRB476#
Record Dates: First submitted 2022-03-15; First posted 2022-04-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Dementia
Keywords: Non-pharmacological interventions; Dementia; Elderly; Randomized Control
MeSH Terms: conditions — Dementia | interventions — Exercise; Cognitive Training; Educational Status

STUDY DESIGN:
Intervention Model Description: * Before the intervention, the research team will record the video for each group:
    * Intervention group: each session comprises (1) 50 min of physical exercise, (2) 20 min of break time or education on dementia and lifestyle habits, and (3) 50 min of cognitive training.
    * Control group: education on dementia and lifestyle habits.
  * Prior to intervening, patients who agree to participate will be screened and evaluated cognitive function, physical function, assessment of Activities of Daily Living, quality of life, depression, anxiety, stress, and sleep quality.
  * We will randomly divide the patients into the intervention-control group at each commune. Each group will attend an "intervention program" once a week within six months.
  * We will evaluate the participants in two groups twice after 3 months and after 6 months of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + cognitive training + education (Experimental): Intervention group: each session comprises (1) 50 min of physical exercise, (2) 20 min of break time or education on dementia and lifestyle habits, and (3) 50 min of cognitive training.
  Interventions: Other: Exercise + cognitive training + education
- Education (Other): Control group: education on dementia and lifestyle habits.
  Interventions: Other: Exercise + cognitive training + education

INTERVENTIONS:
Other: Exercise + cognitive training + education — The research team will record videos for the Intervention group. The intervention procedure includes 3 sections: (1) 50 min of physical exercise, (2) 20 min of break time or lecture on dementia and lifestyle habits, and (3) 50 min of cognitive training. Investigators will be recruited from the National Geriatrics Hospital and trained the technicians for 1 week.
  Prior to intervening, patients who agree to participate will be screened and evaluated cognitive function, physical function, assessment of Activities of Daily Living, quality of life, depression, anxiety, stress, and sleep quality.
  Technicians will record every training session, monitor participants' health, and ensure that those in the intervention group do the exercises correctly.
  We will evaluate the participants in the group after 3 months and after 6 months of intervention.

SUMMARY:
This is a randomized controlled intervention aimed at improving cognitive decline in patients with dementia. The program includes exercise, cognitive training, and dementia education. The output index is expected to be an improvement in cognition, accompanied by an improvement in fitness, sleep quality, reduction in depression levels, and an improvement in quality of life. This is a program that is expected to be effective, inexpensive, easy to apply and does not require high expertise. A total of 50 dementia patients diagnosed and managed by the National Geriatric Hospital, Hai Duong Province General Hospital will be included in the study for 6 months. Patients were randomly assigned to an intervention group and received a program of physical exercise, cognitive training, dementia lecture, and long-term follow-up, or entered a control group to hear a lecture. about dementia. Cognition and fitness will be assessed after follow-up at 0, 3, and 6 months. This work is sponsored by Vingroup Joint Stock Company and supported by domestic Masters/Ph.D. The scholarship program of Vingroup Innovation Fund (VINIF), Vingroup Big Data Institute (VINBIGDATA).

DETAILED DESCRIPTION:
Dementia is a syndrome including memory impairment and other cognitive disorders; that interfere with social and/or professional functioning. The number of people with dementia globally is estimated to increase from 25 million in 2000 to 63 million in 2030. In 2016, dementia was the fifth leading cause of death globally, with approximately 2.4 million people, and one of the leading causes of disability and dependency in the elderly. This affects not only people with dementia but also carers, families, communities, and society; thus, it increases the financial burden on the health system. Healthcare costs for dementia amounted to about $800 billion (accounting for 1% of global GDP) in 2015 and are expected to reach $2 trillion by 2030. Study design: Cluster randomized controlled trial

Study location, time, and subject:

* Location: communes of Thanh Mien district and Gia Loc district of Hai Duong province, Vietnam - the exact location of the REACH Project.
* Time: From 1st January 2021 to 12th December 2022. The investigators started the intervention 6 months after the end of the care capacity-building arm of the REACH project.
* Participants: elderly who are diagnosed with mild and moderate dementia from the aim 1

  * Inclusive criteria: (1) elderly (aged 60 years or above) who are living in Thanh Mien district and Gia Loc district of Hai Duong province; (2) Diagnosed with very mild, mild, and moderate dementia by the Clinical Dementia Assessment (CDR) Questionnaire, corresponding to CDR = 0.5, CDR = 1 and CDR = 2.
  * Exclusive criteria: (1) Not physically fit to participate in physical exercises; (2) Having cardiovascular diseases.

Sample size and sampling process:

* Using the formula for the difference between the 2 ratios, the expected sample size is 25 people in the intervention group and 25 people in the control group.
* Sampling process: randomized cluster sampling

  * Based on the list of patients with dementia diagnosed by a specialist in the initial investigation, The investigators will divide the patients into clusters (communal units) according to where they live.
  * At each research unit (commune), The investigators will randomly divide patients into 2 groups: intervention and control.

Study variables and instruments:

* Outcome variable: The prevalence of mild and moderate dementia pre-and post-intervention are assessed by the Clinical Dementia Assessment (CDR) Questionnaire in Vietnamese
* Independent variables: Daily activity level is assessed using a set of ADLs questionnaires (activities of daily living); Sleep quality according to the PSQI (The Pittsburgh Sleep Quality Index PITTSBURGH); Geriatric depression level according to Geriatric Depression Scale 15 (Geriatric Depression Scale-15); Quality of life according to the Vietnam Quality of Life Scale EQ-5D-5L (European Quality of Life).

Study process:

* The investigators will apply the intervention content based on prior valid evidence by the author "Minoru Kouzuk et al".
* Before the intervention, the research team will record the video for each group:

  * Intervention group: each session comprises (1) 50 min of physical exercise, (2) 20 min of break time or education on dementia and lifestyle habits, and (3) 50 min of cognitive training.
  * Control group: education on dementia and lifestyle habits.
* The research team will recruit and train the technicians at the National Geriatrics Hospital within 1 week.
* Prior to intervening, patients who agree to participate will be screened and evaluated for cognitive function, physical function, assessment of Activities of Daily Living, quality of life, depression, anxiety, stress, and sleep quality.
* The investigators will randomly divide the patients into the intervention-control group at each commune. Each group will attend an "intervention program" once a week for six months. Technicians will record every training session, monitor participants' health, and ensure that those in the intervention group do the exercises correctly.
* The investigators will evaluate the participants in two groups twice after 3 months and after 6 months of intervention.

Data analysis plan and power

* Data entry: The investigators use Kobotoolbox for data entry and management. The investigators use STATA 16.1 and R to clean, process, and analyze data.
* Qualitative variables are calculated by frequency and percentage. The investigators use Fisher Exact Test to determine the differences for qualitative variables and logistic regression to assess the association between outcome and independent variables with odds ratios (OR) and 95% Confidence Interval (95%CI).

ELIGIBILITY:
Inclusion Criteria:

* Elderly (aged 60 years or above).
* Living in Thanh Mien district and Gia Loc district of Hai Duong province.
* Diagnosed with very mild, mild and moderate dementia by the Clinical Dementia Assessment (CDR) Questionnaire, corresponding to CDR = 0.5, CDR = 1 and CDR = 2.

Exclusion Criteria:

* Not physically fit to participate in physical exercises.
* Having cardiovascular diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Changes from Clinical Dementia Rating Questionnaire at 3, and 6 months | Baseline, 3, and 6 months post intervention
  The questionnaire consists of 2 parts: Part 1 is for information providers (relatives/carers), part 2 is for patients, comparing the information provided to evaluate sixaspects, including Memory, Force Orientation, Evaluation - problem-solving, Social activities, Housework - hobbies and Self-care. The study will stimulate both the component scores and the total scores for the dementia grade. The sensitivity of the CDR was 93.6%, a specificity of 100%1. The CDR scale is divided into 5 levels: 0 (No Dementia), 0.5 (Very Mild Dementia), 1 (Mild Dementia), 2 (Moderate Dementia), 3 (Severe dementia).The higher the score, the more severe the dementia

SECONDARY OUTCOMES:
Changes from International Physical Activity Questionnaire - Short Form at 3, and 6 months | Baseline, 3, and 6 months post intervention
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) has been recommended as a cost-effective method to assess physical activity. Only values of 10 or more minutes of activity will be included in the calculation of summary scores. The rationale is that the scientific evidence indicates that episodes or bouts of at least 10 minutes are required to achieve health benefits. This rule is to exclude data that are unreasonably high; these data are to be considered outliers and thus are excluded from the analysis. All Walking, Moderate, and Vigorous time variables that total at least or greater than 16 hours should be excluded from the analysis. The IPAQ-SF scale is divided into 3 levels: Low physical activity, moderate physical activity, and High physical activity. A higher score corresponds to a higher level of physical activity.
Changes from Pittsburgh sleep quality index at 3, and 6 months | Baseline, 3, and 6 months post intervention
  The Pittsburgh sleep quality index (PSQI) was designed as a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time. It includes seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a total score that can range from 0 to 21. A total score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality
Changes from Geriatric Depression Scale-15 at 3, and 6 months | Baseline, 3, and 6 months post intervention
  Geriatric Depression Scale-15 was designed as a self-assessment questionnaire to assess depression in the elderly. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression and 12-15 indicate severe depression. The higher the score, the more severe the depression.
Changes from EuroQoL-5 dimensions-5 levels at 3, and 6 months | Baseline, 3, and 6 months post intervention
  The EQ-5D-5L questionnaire was used to measure the QoL, standardized and applied in Vietnam with Cronbach's alpha = 0.8.The descriptive system contains five dimensions (Mobility, Self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression), which have five levels of response: from no problems (code 1) to extreme problems (code 5). Synthesizing evaluations in 5 different aspects can bring quality of life of respondents. Wallet for example if all 5 aspects are evaluated as no problem, the respondent's health status is 11111. Each health status health corresponds to a composite index defined by international standards for assessing QoL (values from 0 to 1 with 0 representing the worst quality and 1 being the best possible quality). The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam